CLINICAL TRIAL: NCT01349504
Title: Adherence to Mesalamine Profile for Patients With Inflammatory Bowel Disease
Status: Completed | Type: Observational
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Shire (Industry)
Responsible Party: Principal Investigator, Alan C. Moss, Assistant Professor of Medicine, Beth Israel Deaconess Medical Center
Other Study IDs: 2011-P-000067/1
Record Dates: First submitted 2011-04-25; First posted 2011-05-06 (Estimated); Last update posted 2013-08-19 (Estimated); Status verified 2013-08

CONDITIONS: Ulcerative Colitis; Crohn's Disease
MeSH Terms: conditions — Colitis, Ulcerative; Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Mesalmine

SUMMARY:
Hypothesis:

Mesalamine is commonly used to induce and maintain remission in patients with Inflammatory Bowel Disease (IBD). Behavioral and psycho-social barriers to mesalamine adherence exist in patients with IBD. These factors can be identified using qualitative testing in order to develop a validated instrument to measure the "adherence profile" of an individual patient, and design appropriate behavioral interventions to reduce non-adherence.

Objectives:

To test a novel interview instrument that determines the medication adherence profile of patients with IBD prescribed mesalamine by correlating with objective measures of adherence

DETAILED DESCRIPTION:
Specific Aims:

1. To test a novel interview instrument to classify patients into "adherence profiles"
2. To validate this instrument with quantitative scores of mesalamine adherence and objective testing.

Study Design Rationale:

Qualitative research design and prospective validation

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (age >18)
* Diagnosis of IBD (confirmed by endoscopy and histology) > 3 months
* In clinical remission (based on Simple Colitis Activity Index score <2.5)
* On mesalamine compound for maintenance of remission
* Stable mesalamine dose for 1 month

Exclusion Criteria:

* Not receiving primary GI care at BIDMC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients taking mesalamine for maintenance of remission of ulcerative colitis
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2011-04; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Correlation between Adherence to Mesalamine Profile scores and medication adherence as measured by pharmacy refill data | 12 months
  Participant's adherence behaviour will be measured using a behavioral profile questionnaire, and both the total score, and each individual sub-score, correlated with medication adherence as measured using pharmacy refill rates

SECONDARY OUTCOMES:
Self-Reported Adherence (Moriskey Medication Adherence Scale (MMAS) 8 score >6) | 12 months
  Validated measure of reported medication adherence
Spot Urinary 5-ASA | 12 months
  Urine salicylic acid and 5-ASA levels will be measured in participants
Short Inflammatory Bowel Disease Questionnaire | 12 months
  Validated measure of Quality-of-Life for patients with IBD
Pharmacy Refill Rates | 12 months
  Mesalamine refill rates will be captured from patiernts' pharmacies

CONTACTS AND LOCATIONS:
Overall Officials: Alan Moss, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Moss AC, Lillis Y, Edwards George JB, Choudhry NK, Berg AH, Cheifetz AS, Horowitz G, Leffler DA. Attitudes to mesalamine questionnaire: a novel tool to predict mesalamine nonadherence in patients with IBD. Am J Gastroenterol. 2014 Dec;109(12):1850-5. doi: 10.1038/ajg.2014.158. Epub 2014 Jun 10. PMID 24913040
- See also: Related Info — http://www.bidmc.org/CentersandDepartments/Departments/DigestiveDiseaseCenter/InflammatoryBowelDiseaseProgram.aspx